CLINICAL TRIAL: NCT04489797
Title: A Phase I, Open-label, Randomized, Single-dose Study of Acalabrutinib in Healthy Subjects to Evaluate the Effect of Proton-pump Inhibitor (Rabeprazole) on Acalabrutinib Capsule When Administered Orally With COCA-COLA
Brief Title: A Study to Evaluate Effects of Proton-pump Inhibitor on Acalabrutinib Capsule When Administered Orally With COCA-COLA in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D822FC00008
Record Dates: First submitted 2020-07-27; First posted 2020-07-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Infectious Disease
Keywords: Pharmacokinetics; Bioavailability
MeSH Terms: conditions — Communicable Diseases | interventions — acalabrutinib; Rabeprazole

STUDY DESIGN:
Intervention Model Description: This is open-label, randomized, single-dose study. The participants will be divided in 2 treatment arms as follows:
  1. Arm A (only acalabrutinib)
  2. Arm B (acalabrutinib + rabeprazole)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will receive single oral dose of acalabrutinib capsule with 100 mL of water.
  Interventions: Drug: Acalabrutinib
- Arm B (Experimental): Participants will receive single oral dose of acalabrutinib capsule taken with 100 mL of COCA-COLA along with 20 mg rabeprazole.
  Interventions: Drug: Acalabrutinib; Drug: Rabeprazole

INTERVENTIONS:
Drug: Acalabrutinib — Participants will receive single oral dose of acalabrutinib on day 1 as per the arms they are randomized.
Drug: Rabeprazole — Participants will receive twice daily oral dose of 20 mg rabeprazole on days -3, -2, and -1.
  Arms: Arm B

SUMMARY:
This study is being conducted to support the clinical development of acalabrutinib in participants who need treatment with proton pump inhibitors while taking acalabrutinib.

DETAILED DESCRIPTION:
This is an open-label, single-center, randomized study in healthy participants to evaluate the effect of proton-pump inhibitors (rabeprazole; PPI) on acalabrutinib 100-mg capsule dosed orally with COCA-COLA. Participants will receive a single dose of acalabrutinib alone or with rabeprazole, and pharmacokinetic (PK), safety and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Male participants and their female partners/spouses must adhere to the contraception methods.
* Female participants must have a negative pregnancy test at screening, must not be lactating, and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  * Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and follicle stimulating hormone levels in the postmenopausal range.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not bilateral tubal ligation.
* Have a body mass index between 18.5 and 30 kg/m^2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive, at screening.
* Understands the study procedures in the informed consent form and willing and able to comply with the protocol.

Exclusion Criteria:

* History or presence of any clinically significant disease (including active coronavirus disease 2019 infection).
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 30 days of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormalities in hematology, coagulation, clinical chemistry, or urinalysis results, at screening defined as:

  * Hemoglobin less than lower limit of normal.
  * Serum alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase or serum bilirubin (total and direct) > 1.5 upper limit of normal.
* Any clinically significant abnormal findings in vital signs at screening (eg, systolic blood pressure [BP] < 90 mmHg or ≥ 140 mmHg; diastolic BP < 50 mmHg or ≥ 90 mmHg; pulse < 50 or > 90 bpm).
* Any clinically significant abnormalities on standard 12-lead electrocardiogram at screening.
* Any positive result on screening for serum Hepatitis B surface antigen, hepatitis B, hepatitis C, and Human immunodeficiency virus antibody.
* Has received a new chemical entity within 90 days of the first administration of IMP in this study. The period of exclusion begins 90 days after the final dose or 30 days after the last visit whichever is the longest.
* Plasma donation within 30 days of screening or any blood donation/loss more than 500 mL during the 90 days prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to acalabrutinib or rabeprazole.
* Current smokers or those who have smoked or used nicotine products within the 90 days prior to screening.
* Positive screen for drugs of abuse or cotinine at screening.
* Treatment with a strong cytochrome P450 3A (CYP3A) inhibitor (within 14 days before first administration of IMP) or strong CYP3A inducer (within 28 days before first administration of IMP).
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 14 days prior to the first administration of IMP or longer if the medication has a long half-life. Hormonal replacement therapy will not be allowed.
* Known or suspected history of alcohol or drug abuse, or excessive intake of alcohol.
* Excessive intake of caffeine-containing drinks or food or would likely be unable to refrain from the use of caffeine-containing beverages during in-house stay at the Clinical Unit.
* Involvement of any AstraZeneca, Acerta Pharma, Parexel or study site employee or their close relatives.
* Judgment by the Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Participants who cannot communicate reliably with the Investigator.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Inability to swallow acalabrutinib capsules.
* Evidence of ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections). Note: Participants with localized cutaneous fungal infections are eligible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUCinf) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on Day 1, and 24 hours post-dose on Day 2
  Assessment of AUCinf for acalabrutinib and ACP-5862 (metabolite of acalabrutinib) following administration of capsule with and without rabeprazole.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on Day 1, and 24 hours post-dose on Day 2
  Assessment of AUClast for acalabrutinib and ACP-5862 following administration of capsule with and without rabeprazole.
Maximum observed plasma concentration (Cmax) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on Day 1, and 24 hours post-dose on Day 2
  Assessment of Cmax for acalabrutinib and ACP-5862 following administration of capsule with and without rabeprazole.

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events | From screening until Follow-up visit (Upto 5 to 6 Weeks)
  Assessment of the safety and tolerability of acalabrutinib capsule when administered with COCA-COLA and rabeprazole.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Winkle, MD FACP FACG CPI, Principal Investigator — Anaheim Clinical Trials
Locations (1):
- Research Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home